CLINICAL TRIAL: NCT06182332
Title: Piloting an Artificial Intelligence Algorithm Used to Identify Patients in Need of Outpatient (or Ambulatory) Palliative Care in an Oncology Population
Brief Title: An Artificial Intelligence Algorithm for Identifying Gynecologic Cancer Patients in Need of Outpatient Palliative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 23-008371; NCI-2023-09943 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-008371 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2023-12-08; First posted 2023-12-26 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Advanced Malignant Female Reproductive System Neoplasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Screening (AI algorithm) (Experimental): Patients' medical records are reviewed for consideration of palliative care consult using AI algorithm QW for 6 months.
  Interventions: Other: Electronic Health Record Review; Other: Internet-Based Intervention

INTERVENTIONS:
Other: Electronic Health Record Review — Undergo medical record review
Other: Internet-Based Intervention — Use AI algorithm

SUMMARY:
This clinical trial tests an artificial intelligence (AI) algorithm for its ability to identify patients who may benefit from a palliative care consult for gynecologic cancer that has spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced). A significant delay in referral to palliative care often occurs among patients with cancer. This delay can lead to poorer symptom management, decreased quality of life, and care that does not align with patient goals or values. AI algorithms are computer programs that use step-by-step procedures to solve a problem. In this trial, an AI algorithm is applied to patients' medical records in order to identify patients with a high burden of disease. Information gathered from this study may help researchers learn whether this AI algorithm is useful for identifying patients who could benefit from outpatient palliative care consultation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To pilot an oncology risk prediction model to identify patients who may benefit from outpatient palliative care consultation to improve symptom management and goal-concordant care in this population.

OUTLINE:

Patients' medical records are reviewed for consideration of palliative care consult using AI algorithm once a week (QW) for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient in Enhanced, Electronic health record (EHR)-facilitated Cancer Symptom Control (E2C2) with a diagnosis of advanced gynecologic malignancy (International Classification of Diseases [ICD] codes C51 through C58)
* Weekly the reviewers will select patients by looking at patients in sorted order starting with the highest score and proceeding down the list and evaluating each patient for exclusion criteria

Exclusion Criteria:

* Patients that have been seen by palliative care will be excluded for 75 days
* Patients under the age of 18 years
* Patients currently enrolled with hospice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2023-12-11 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Timely identification for need of palliative care | Up to 6 months
  Will be measured as time to the electronic record of consult by the palliative care team in the outpatient setting.

SECONDARY OUTCOMES:
Number of palliative care consultations | Up to 6 months
  Number of palliative care consultations will be assessed as the number of participants who receive palliative care consultations.
Number of advanced care planning notes documented in the electronic health record | Up to 6 months
  Participant electronic health records will be reviewed for the number of advanced care planning notes listed.
Number of billing codes International Classification of Diseases, 10th Revision for palliative care | Up to 6 months
  Participant electronic health records will be reviewed for the number of International Classification of Diseases, 10th Revision (ICD-10) billing codes for palliative care.
Positive predictive value of screened patients | Up to 6 months
  Will be assessed as the number of patients identified by Artificial Intelligence algorithm who actually received palliative care consultation.
Performance metrics on reviewer/oncologist handoff | Up to 6 months
  Will be assessed by agreement statistics and descriptive statistics on time between oncology contact and oncology response.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel D. Havyer, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials